CLINICAL TRIAL: NCT06930001
Title: Effect of Etamine Processing on Midwifery Students' Episiotomy Repair Application Ability, Perceived Stress and Learning Attitude: Randomized Controlled Study
Brief Title: Etamine Processing on Episiotomy Repair Skills, Stress and Learning Attitudes in Midwifery Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Şeyma Demir, MsC, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1234567891
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Episiotomy Repair Skills; Learning Attitude
Keywords: perceived stress; midwifery student
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etamine Application Group /Intervention (Experimental): Before the intervention, students in the intervention group will complete the Informed Consent Form, Personal Information Form, Perceived Stress Scale, and Attitudes Towards Learning Scale (pre-test). In the first week, a 45-minute etamine training will be provided individually by the scholarship holder (Şeyma Demir) in the clinical skills lab. Basic techniques will be taught and students will apply a simple pattern. Environmental conditions (21℃) and student comfort will be ensured, and the room will be restricted during practice. One week later, students will continue etamine practice for three weeks, 45 minutes per week. In the fifth week, the project manager will deliver episiotomy training (2 hours theory, 4 hours practice), followed by assessment in the clinical lab using the Episiotomy Repair Skill Form (post-test). Final evaluations will include the Perceived Stress Scale and the Attitudes Towards Learning Scale (post-test).
  Interventions: Other: Etamine Application Group /Intervention
- Control (No Intervention): Control group students will receive the same episiotomy training (2 hrs theory, 4 hrs practice) as the intervention group, without the additional etamine application. They will complete the Informed Consent Form, Personal Information Form, Perceived Stress Scale, and Attitudes Towards Learning Scale (pre-test) during the first meeting. Measurement conditions (21℃ room temperature, restricted access) will be standardized to ensure comfort and reduce bias. Five weeks later, episiotomy training will be delivered by the project manager, followed by observational assessment using the Episiotomy Repair Skill Form (post-test). Final evaluations will also include the Perceived Stress Scale and the Attitudes Towards Learning Scale. After the study, etamine training will be optionally offered to the control group to ensure equal skill opportunities.

INTERVENTIONS:
Other: Etamine Application Group /Intervention — Before the intervention, students in the intervention group will complete the Informed Consent Form, Personal Information Form, Perceived Stress Scale, and Attitudes Towards Learning Scale (pre-test). In the first week, a 45-minute etamine training (history, tools, basic techniques) will be given individually by the scholarship holder (Şeyma Demir). Techniques such as threading, knotting, and cross-stitching will be taught, and students will apply a simple pattern, correcting mistakes. Room conditions (21℃) and student comfort will be ensured, with restricted access. One week later, students will practice weekly for 3 weeks (45 minutes each) using the Etamine starter set. In week five, the project manager will provide 2 hours of theory and 4 hours of practical episiotomy training. Students will then be assessed with the Episiotomy Repair Skill Form (post-test). Final evaluations will include the Perceived Stress Scale and Attitudes Towards Learning Scale (post-test).
  Arms: Etamine Application Group /Intervention

SUMMARY:
Research Hypotheses H1: Midwifery students who practice Etamine have higher episiotomy repair skills than those who do not.

H2: Midwifery students who practice Etamine have lower perceived stress levels than those who do not.

H3: Midwifery students who practice Etamine have higher learning attitudes than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study include students who are willing to participate in the study and who do not have any learning or working experience related to episiotomy repair.

Exclusion Criteria:

* Students with diagnosable diseases affecting their learning ability, those who have had accidents during the training and assessment sessions, and foreign nationals will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As midwifery students must be female, only women are accepted in Türkiye.
Enrollment: 104 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Episiotomy Repair Skill Form | Fifth week after the start of the application
  The form, which was developed by the researcher by scanning the literature and obtaining expert opinions, consists of 16 questions. It will be evaluated under four headings. It consists of "Selection and use of suture material (3 questions)", "Suture Technique and Application (8 questions)", "Equal and Proper Placement of Sutures (2 questions)", "Aesthetic and Functional Results (3 questions)". The steps in the skill form were examined by midwifery faculty members who are experts in the field and finalized. The evaluation form includes the following options: "1. Needs improvement: The step is not applied at all, applied incorrectly or not applied in order, 2. Sufficient: The step is applied correctly and in order, but there are deficiencies and/or the help of the trainer is needed, 3. Mastered: The step is applied correctly and in order without pausing and needing help." High scores obtained from the form indicate good skill.
Perceived Stress Scale | pre-intervention
  The Perceived Stress Scale (PSS-10), developed by Cohen et al. (1983) and adapted to Turkish by Kaya et al. (2019), consists of 10 items rated on a five-point Likert scale (0-4). Items 4, 5, 7, and 8 are reverse-scored. Scores of 0-13 indicate low, 14-26 moderate, and 27-40 high stress. Cronbach's alpha for self-efficacy and helplessness subscales were 0.68 and 0.85, respectively. The scale was used to assess how stress in the lab setting affects students' skill performance and reflects clinical stress. The lab is a preparatory stage for clinical practice, making stress measurement here significant. Literature shows that lab stress can impact students' skills (Duffy et al., 2021), and tasks requiring fine motor skills like etamine may also influence stress in competitive environments (Ferrara, 2022). Therefore, the PSS will evaluate both lab stress and etamine's impact, contributing valuable insights into skill performance and preparedness.
Attitude Scale Towards Learning | pre-intervention
  The scale was developed by Kara (2010) to measure students' attitudes towards learning. It includes 40 items and four sub-dimensions: Nature of Learning (7 items), Anxiety About Learning (13 items), Expectations About Learning (9 items), and Openness to Learning (11 items). It uses a 5-point Likert scale: 1 (Strongly Disagree) to 5 (Strongly Agree). Subscale score ranges are: Nature of Learning (7-35), Anxiety (13-65), Expectations (9-45), and Openness (11-55). The scale provides insights into how students perceive and approach learning. Cronbach's alpha was calculated as 0.73, indicating acceptable reliability (Kara, 2010). It is suitable for assessing both positive and negative attitudes related to the learning process in educational research.

SECONDARY OUTCOMES:
Perceived Stress Scale | Fifth week after the start of the application
  The Perceived Stress Scale (PSS-10), developed by Cohen et al. (1983) and adapted to Turkish by Kaya et al. (2019), consists of 10 items rated on a five-point Likert scale (0-4). Items 4, 5, 7, and 8 are reverse-scored. Scores of 0-13 indicate low, 14-26 moderate, and 27-40 high stress. Cronbach's alpha for self-efficacy and helplessness subscales were 0.68 and 0.85, respectively. The scale was used to assess how stress in the lab setting affects students' skill performance and reflects clinical stress. The lab is a preparatory stage for clinical practice, making stress measurement here significant. Literature shows that lab stress can impact students' skills (Duffy et al., 2021), and tasks requiring fine motor skills like etamine may also influence stress in competitive environments (Ferrara, 2022). Therefore, the PSS will evaluate both lab stress and etamine's impact, contributing valuable insights into skill performance and preparedness.
Attitude Scale Towards Learning | Fifth week after the start of the application
  The scale was developed by Kara (2010) to measure students' attitudes towards learning. It includes 40 items and four sub-dimensions: Nature of Learning (7 items), Anxiety About Learning (13 items), Expectations About Learning (9 items), and Openness to Learning (11 items). It uses a 5-point Likert scale: 1 (Strongly Disagree) to 5 (Strongly Agree). Subscale score ranges are: Nature of Learning (7-35), Anxiety (13-65), Expectations (9-45), and Openness (11-55). The scale provides insights into how students perceive and approach learning. Cronbach's alpha was calculated as 0.73, indicating acceptable reliability (Kara, 2010). It is suitable for assessing both positive and negative attitudes related to the learning process in educational research.

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting in April 2024
Access Criteria: The IPD will be shared with principal researchers.